CLINICAL TRIAL: NCT03262688
Title: A Multicenter, Randomized, Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Analgesic Effect of the INL-001 Bupivacaine Hydrochloride (HCl) Collagen-Matrix Implant in Children 2 to <17 Years of Age Following Open Inguinal Hernia Repair
Brief Title: Safety, Tolerability, PK, and Analgesic Effect of INL-001 in Children Following Open Inguinal Hernia Repair
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INN-CB-020
Record Dates: First submitted 2017-08-21; First posted 2017-08-25 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Inguinal Hernia; Postoperative Pain
Keywords: INL-001; Bupivacaine; Collagen; Children; Pediatric; Inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Randomized, controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant, legal guardian and study personnel involved in the assessment of efficacy and safety are blinded to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INL-001 (Experimental): Bupivacaine HCl collagen-matrix implant
  Interventions: Drug: Bupivacaine HCl collagen-matrix implant
- Infiltration (Active Comparator): Bupivacaine HCl infiltration
  Interventions: Drug: Bupivacaine HCl infiltration

INTERVENTIONS:
Drug: Bupivacaine HCl collagen-matrix implant — Placement of the bupivacaine collagen-matrix in the surgical site
  Other Names: Xaracoll
  Arms: INL-001
Drug: Bupivacaine HCl infiltration — Infiltration of the surgical site
  Other Names: Marcaine
  Arms: Infiltration

SUMMARY:
A multicenter, single-dose study in children 12 to <17 years of age, 6 to <12 years of age, and 2 to <6 years of age who are scheduled for elective open inguinal hernia repair. Enrollment in this study will start with the oldest age group (12 to <17 years) and will continue in a stepwise fashion until appropriate doses are established for all 3 pediatric age groups (12 to <17 years, 6 to <12 years, 2 to <6 years).

DETAILED DESCRIPTION:
This is a multicenter, single-dose study in children 12 to <17 years of age, 6 to <12 years of age, and 2 to <6 years of age who are scheduled for elective open inguinal hernia repair. Within 21 days of surgery, eligible subjects will be screened and have routine clinical laboratory testing and an electrocardiogram performed. Subjects will then undergo an open inguinal hernia repair under general anesthesia according to the investigator's standard surgical practice on day 1. Enrollment in this study will start with the oldest age group (12 to <17 years) and will continue in a stepwise fashion until appropriate doses are established for all 3 pediatric age groups. Within each age group, the study will be conducted in 3 parts.

Children in each age group who are randomized to INL-001 will receive approximately less than or equal to 2.5 mg/kg of INL-001. Study drug will be administered prior to wound closure. The INL-001 implant will be cut before placement into the surgical site using sterile technique. Children randomized to 0.25% bupivacaine HCl injection will receive 2.5 mg/kg according to standard practice.

After completion of the surgical procedure, all subjects will remain in the post-anesthesia care unit for at least 3 hours and will be continuously monitored for safety. At the discretion of the investigator, subjects may receive rescue medication (opioid or nonopioid) upon request for the management of breakthrough pain and may receive an antiemetic for the management of nausea or vomiting. After the initial 3-hour period, subjects who are deemed stable may be discharged to the hospital ward. Subjects will remain housed in the hospital ward for at least 48 hours. Blood samples will be collected for pharmacokinetic analysis from a subset of 8 children in each age group after INL-001 is implanted.

ELIGIBILITY:
Inclusion Criteria:

* Be a male or female 2 to <17 years of age.
* Be eligible for an elective open inguinal hernia repair that will be performed according to standard surgical technique under general anesthesia.
* Be premenarche or have a serum confirmed negative pregnancy test at screening and a negative urine pregnancy test before surgery on day 1, if an adolescent female of childbearing potential.
* Be willing and able to cooperate with all the requirements of the study.
* Be able to speak and understand English or Spanish.
* Have a legally authorized representative (eg, parent, guardian) who is able to read, speak, and understand English or Spanish and who will voluntarily sign and date a parental permission/informed consent form that is approved by the Institutional Review Board/Independent Ethics Committee/Human Research Ethics Committee (IRB/IEC/HREC).
* Be willing to sign an assent (if appropriate dependent upon the child's age, understanding, and IRB requirements), before the conduct of any study procedure.

Exclusion Criteria:

* Has a known hypersensitivity to amide local anesthetics, bovine products, or to inactive ingredients of the study drugs.
* Requires any additional surgical procedures, either related or unrelated to the scheduled surgery (ie, open inguinal hernia surgery), during the same hospitalization.
* Requires epidural or spinal blockade perioperatively.
* Is required to receive neuraxial (spinal or epidural) opioid analgesics during the study.
* Has undergone major surgery within 3 months of the scheduled surgery or plans to undergo another surgical procedure within the 30-day postoperative period.
* Has known or suspected history of drug abuse or misuse or evidence of tolerance or physical dependency on opioid analgesics or sedative-hypnotic medications.
* Has participated in a clinical trial (investigational or marketed product) within 30 days before surgery.
* Has any clinically significant medical history or condition (eg, unstable cardiac, neurological, immunological, renal, hepatic, or hematological disease or any other condition) that in the opinion of the investigator, substantially increases the risk associated with the subject's participation in the protocol or compromises the scientific objectives of the study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Estimated)
Dates: Start 2017-06-16 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 30 days
  Possibly related to bupivacaine toxicity
Blood pressure (systolic/diastolic) | Starting at Time 0 and continuing for 3 hours and then 5, 8, 12, 24, 36, and 48 hours after Time 0
  Signs/symptoms of bupivacaine toxicity
Heart rate | Continuously from Time 0 through 3 hours, and then 5, 8, 12, 24, 36, and 48 hours after Time 0
  Signs/symptoms of bupivacaine toxicity
Respiratory rate | Continuously from Time 0 through 3 hours, and then 5, 8, 12, 24, 36, and 48 hours after Time 0
  Signs/symptoms of bupivacaine toxicity
Body temperature | Through Day 30
  Signs/symptoms of bupivacaine toxicity
12-lead ECG | 1 day at screening
  Screening only
3-lead ECG | Starting at Time 0 and continuing for at least 3 hours
  Signs/symptoms of bupivacaine toxicity
Oxygen saturation levels | Starting at Time 0 and continuing for at least 3 hours
  Pulse oximetry
Clinical laboratory testing | 1 day at screening
  Collection of blood and urine samples
Wound healing assessments | Assessment on Day 1 through Day 3; follow-up evaluations on Days 7, 15 and 30
  Inspection of surgical wound site for signs of wound infection and dehiscence.
Nausea | 1, 2, 4, 6, 12, 24, 36, and 48 hours after Time 0
  Measured using a categorical scoring system (none = 0, mild = 1, moderate = 2, and severe = 3). Nausea scores will also be recorded immediately before the use of rescue antiemetics
Sedation | 1, 2, 4, 6, 12, 24, 36, and 48 hours after Time 0
  Sedation scores: awake and alert = 0, quietly awake = 1, asleep but easily roused = 2, and deep sleep = 3.

SECONDARY OUTCOMES:
Cmax | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hour time points after Time 0.
  Maximum observed plasma concentration
AUC0-last | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hour time points after Time 0
  Area under the plasma concentration time curve from Time zero to last quantifiable plasma concentration
AUC0-∞ | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hour time points after Time 0
  Area under the plasma concentration time curve from Time zero to extrapolated through infinity
Tmax | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hour time points after Time 0
  Time to maximum obserbved plasma concentration
t1/2 | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 18, 24, 36, and 48 hour time points after Time 0
  Apparent first-order terminal elimination half-life
Pain intensity | 1, 2, 4, 6, 12, 24, 36, and 48 hours after Time 0
  Assessed using an 11-point NRS (for children 12 to <17 years of age), a FACES pain severity scale (children 4 through <12 years of age), or FLACC (children 2 and 3 years of age) immediately before the child receives any parenteral or oral rescue medication for breakthrough pain

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Niebler, DO, Study Director — Innocoll
Locations (11):
- United States (11):
  - Alliance Research Centers, Laguna Hills, California
  - Cornerstone Research Institute, Altamonte Springs, Florida
  - Medical Research Center, Miami, Florida
  - Elion & Volhard Pharmaceutical Research (E&V PR), Miami, Florida
  - Children's Hospital of Pittsburgh of UPMC (CHP-UPMC), Pittsburgh, Pennsylvania
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - Plano Surgical Hospital, Plano, Texas
  - Jean Brown Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No